CLINICAL TRIAL: NCT00298272
Title: A Randomized, Double-Blinded, Placebo Controlled Study to Evaluate the Tolerability and Safety of Rituximab When Given in Combination With Methotrexate and Etanercept (Enbrel) or Methotrexate and Adalimumab (Humira) in Subjects With Active Rheumatoid Arthritis
Brief Title: Safety and Tolerability of Rituxan With Methotrexate and Etanercept or Methotrexate and Adalimumab in Patients With Active Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decided to end long term extension phase for business reasons unrelated to safety.
Sponsor: Biogen (Industry)
Collaborators: Hoffmann-La Roche (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 102-RA-201
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Results first posted 2010-11-17 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate; Etanercept; Adalimumab; Methylprednisolone; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double-blind/Open Label Rituximab (Experimental): The double-blind rituximab treatment group received rituximab 500 mg by intravenous (IV) infusion on Day 1 and Day 15. After 24 weeks (primary endpoint completion), participants continued post-treatment follow-up (PTFU) visits through Week 56, and entered a 48-week Safety Follow-Up (SFU). At any time between Week 24 and Week 40 of PTFU, eligible participants could enter the rituximab open label (OL) arm, and "restart" the 56-week treatment/follow-up schedule (rituximab 500 mg by IV infusion on Day 1 and Day 15) prior to the 48-week SFU.
  Prior to rituximab infusion, participants were premedicated with methylprednisolone 100 mg IV. Participants received folate ≥5 mg weekly. Background therapy (stable dose for the duration of the study) included: a tumor necrosis factor (TNF) inhibitor; either etanercept 50 mg subcutaneous injection (SC) weekly or adalimumab 40 mg SC once every 2 weeks; methotrexate (MTX) 15 to 25 mg by mouth or by intramuscular injection (IM) weekly.
  Interventions: Biological: IDEC-C2B8 (rituximab); Drug: Methotrexate; Drug: Etanercept; Drug: Adalimumab; Drug: Methylprednisolone; Dietary Supplement: Folate
- Double-blind Placebo/Open Label Rituximab (Other): The double-blind placebo treatment group received saline solution IV on Day 1 and Day 15. After 24 weeks (primary endpoint completion), participants continued post-treatment follow-up (PTFU) visits through Week 56, and entered a 48-week Safety Follow-Up (SFU). At any time between Week 24 and Week 40 of PTFU, eligible participants could enter the rituximab open label (OL) arm, and "restart" the 56-week treatment/follow-up schedule (rituximab 500 mg by IV infusion on Day 1 and Day 15) prior to the 48-week SFU.
  Prior to each infusion of placebo, participants were premedicated with methylprednisolone 100 mg IV. Participants received folate ≥5 mg weekly. Background therapy (stable dose for the duration of the study) included: a tumor necrosis factor (TNF) inhibitor; either etanercept 50 mg subcutaneous injection (SC) weekly or adalimumab 40 mg SC once every 2 weeks; methotrexate (MTX) 15 to 25 mg by mouth or by intramuscular injection (IM) weekly.
  Interventions: Drug: Placebo; Drug: Methotrexate; Drug: Etanercept; Drug: Adalimumab; Drug: Methylprednisolone; Dietary Supplement: Folate

INTERVENTIONS:
Biological: IDEC-C2B8 (rituximab) — Participants will receive 500 mg rituximab on Day 1 and Day 15
  Other Names: Rituxan
  Arms: Double-blind/Open Label Rituximab
Drug: Placebo — Participants will receive placebo on Day 1 and Day 15
  Arms: Double-blind Placebo/Open Label Rituximab
Drug: Methotrexate — Participants must have been treated with MTX ≥15 mg per week and ≤25 mg per week (dose may have been as low as 10 mg if unable to tolerate higher dose) for at least 12 weeks immediately prior to Day 1, at a stable dose for at least 4 weeks and was continued for the study duration.
Drug: Etanercept — Participants must have been treated with etanercept at 50 mg per week (25 mg twice per week or 50 mg once per week).
  Other Names: Enbrel
Drug: Adalimumab — Participants must have been treated with adalimumab at 40 mg every other week for at least 12 weeks immediately prior to Day 1.
  Other Names: Humira
Drug: Methylprednisolone — Methylprednisolone 100 mg IV was administered by slow infusion to be completed at least 30 minutes prior to each infusion of rituximab or placebo.
Dietary Supplement: Folate — All subjects also received a stable dose of folate (≥5 mg per week).

SUMMARY:
The primary objective of this study was to evaluate the tolerability and safety of rituximab in combination with methotrexate (MTX) and etanercept or adalimumab in participants with active rheumatoid arthritis (RA). The secondary objective was to explore the efficacy of rituximab in combination with MTX and etanercept or adalimumab in participants with active RA.

DETAILED DESCRIPTION:
The study consists of 4 parts: screening, treatment, post-treatment, and safety follow-up. Prior to Day 1, participants were discontinued from all disease-modifying anti-rheumatic drugs (DMARDs) except MTX and etanercept or adalimumab. All participants who met eligibility criteria and were enrolled in the trial were randomized to receive 500 mg rituximab or placebo on Day 1 and Day 15. A subset of 18 participants was enrolled initially and followed through Week 12 for safety. The remaining 42 participants were to be enrolled after the last participant in the subset completed Week 12 and the Data Safety Monitoring Board (DSMB) conducted a safety review and approved enrollment of these additional participants. Participants were dosed on Day 1 and Day 15 and followed for 56 weeks, while remaining on their current dose of MTX and etanercept or adalimumab throughout the study. The primary endpoint was assessed at Week 24.

All participants in double-blind treatment, including those who received placebo or rituximab, who met the open label inclusion/exclusion criteria anytime from Week 24 through Week 40, were eligible to enter the open label retreatment phase. These participants received open label rituximab on Day 1 and Day 15 of the retreatment phase, and were followed monthly until Week 24 then every 2 months until Week 56, while remaining on their current dose of MTX and etanercept or adalimumab throughout the study. Participants received 1 course of open label treatment only.

All participants were required to return for safety follow-up (SFU) assessments at Weeks 4, 12, 24, 36, and 48 after withdrawal or completion of the study. Participants whose peripheral CD20+ B cells remained depleted at the end of the SFU periods for the primary and OL portions of the study entered extended safety follow-up (ESFU). Assessments for ESFU were performed at 12-week intervals until peripheral B-cell levels returned to within normal range or baseline level (whichever was lower).

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent. If required by local law, candidates must also authorize the release and use of protected health information (PHI).
2. Male or female participants, between 18 and 65 years of age, who have a diagnosis of active RA for at least 6 months, diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria for the classification of rheumatoid arthritis (RA).
3. Must have at least 5 tender and 5 swollen joints at Screening and Day 1.
4. Must have been treated with etanercept at 50 mg per week (25 mg twice per week or 50 mg once per week) or adalimumab at 40 mg every other week for at least 12 weeks immediately prior to Day 1.
5. Must have been treated with methotrexate (MTX) greater than or equal to 15 mg per week and less than or equal to 25 mg per week (dose may be as low as 10 mg if unable to tolerate higher dose) for at least 12 weeks immediately prior to Day 1, at a stable dose for at least 4 weeks.
6. Must be willing to receive oral folate.
7. Oral glucocorticoids must not exceed 10 mg per day of prednisone (or equivalent dose) and must have been administered at a stable dose for at least 4 weeks prior to Day 1.
8. Any concomitant non-steroidal antiinflammatory drugs (NSAIDs) must be stable for at least 2 weeks prior to Day 1.
9. For participants of reproductive potential (males and females), use of a reliable means of contraception (e.g., hormonal contraceptive, patch, intrauterine device, physical barrier) throughout study participation.

   Exclusion Criteria:

   Exclusions Related to RA
10. Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis, or Felty's syndrome). Secondary Sjögren's syndrome or secondary limited cutaneous vasculitis with RA is permitted.
11. Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis.
12. History of, or current, inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus [SLE], inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, or any overlap syndrome).
13. Diagnosis of juvenile idiopathic arthritis, also known as juvenile RA, and/or RA before age 16.

    Exclusions Related to General Health
14. Any surgical procedure, including bone/joint surgery/synovectomy (including joint fusion or replacement) within 12 weeks prior to baseline or planned within 24 weeks of randomization.
15. Lack of peripheral venous access.
16. Pregnancy or breast feeding.
17. Significant cardiac or pulmonary disease (including obstructive pulmonary disease).
18. History of chronic heart failure (CHF), SLE-like syndrome, neuropathy or myelitis, optic neuritis, or pancytopenia while on etanercept or adalimumab.
19. Evidence of significant uncontrolled concomitant disease such as, but not limited to, nervous system, renal, hepatic, endocrine, or gastrointestinal disorders which, in the investigator's opinion, would preclude subject participation.
20. Primary or secondary immunodeficiency (history of, or currently active), including known history of human immunodeficiency virus (HIV) infection.
21. Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with IV anti infectives within 4 weeks of Day 1 or completion of oral anti infectives within 2 weeks of Day 1.
22. History of positive purified protein derivative (PPD) not adequately treated.
23. History of deep space/tissue infection (e.g., fasciitis, abscess, osteomyelitis) within 52 weeks of Day 1.
24. History of serious infection or opportunistic infection in the last 2 years (to screen for a chest infection, a chest radiograph will be performed at Screening if one was not performed within 12 weeks prior to Screening).
25. History of seizures.
26. History of cancer, including solid tumors, hematologic malignancies, and carcinoma in situ (except basal cell and squamous cell carcinoma of the skin that have been excised and cured).
27. Any neurological (congenital or acquired), vascular, or systemic disorder that might affect any of the efficacy assessments, in particular, joint pain and swelling (e.g., Parkinsons disease, cerebral palsy, diabetic neuropathy).
28. Currently active alcohol or drug abuse or history of alcohol or drug abuse (as determined by the Investigator) within 1 year prior to Day 1.

    Exclusions Related to Medications
29. History of a severe allergic or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of rituximab or to murine proteins.
30. Previous treatment with an anti alpha 4 integrin agent or costimulation modulator.
31. Concurrent treatment with any biologic agent other than etanercept or adalimumab, or disease-modifying anti-rheumatic drug (DMARD) other than MTX. Treatment with any biologic or DMARD except etanercept or adalimumab, and MTX must be discontinued 14 days prior to baseline, except for the following: azathioprine for 28 days; leflunomide for 8 weeks (or 14 days after 11 days of standard cholestyramine or activated charcoal washout).
32. Previous treatment with any cell depleting therapies, including investigational agents (e.g., Campath [alemtuzumab], anti-CD4, anti-CD5, anti-CD3, anti-CD19, anti CD11a, anti-CD22, B lymphocyte stimulator/B-cell activating factor [BLys/BAFF], and anti-CD20).
33. Treatment with another investigational drug within 4 weeks prior to Day 1 or 5 half lives of the investigational drug (whichever is the longer).
34. Receipt of a live/attenuated vaccine within 4 weeks prior to Day 1.
35. Intra-articular or parenteral glucocorticoids within 4 weeks prior to Day 1.
36. Intolerance or contraindications to IV glucocorticoids.

    Exclusions Related to Laboratory Findings
37. For women of childbearing potential, a positive serum pregnancy test at screening and/or a positive urine pregnancy test on Day 1.
38. Positive hepatitis B surface antigen (HBsAg).
39. Positive hepatitis B core antibody (HBcAb) associated with positive hepatitis B viral DNA (HBV DNA).
40. Positive hepatitis C antibody.
41. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times upper limit of normal.
42. Hemoglobin <8.0 g/dL.
43. Levels of immunoglobulin G (IgG) and/or immunoglobulin M (IgM) below 5.0 and 0.4 mg/mL, respectively.
44. Absolute neutrophil count (ANC) <1500/mL.

    Miscellaneous Exclusions
45. Current enrollment in any other investigational or other drug study.
46. Treatment with IV Gamma Globulin or the Prosorba® Column within 6 months of the Screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- United States (18):
  - Research Site, Huntsville, Alabama
  - Research Site, Paradise Valley, Arizona
  - Research Site, Palm Desert, California
  - Research Site, Jupiter, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Boise, Idaho
  - Research Site, Kalamazoo, Michigan
  - Research Site, St Louis, Missouri
  - Research site, Chardon, Ohio
  - Research Site, Mayfield Village, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Burlington, Vermont

REFERENCES:
- [Result] Greenwald MW, Shergy WJ, Kaine JL, Sweetser MT, Gilder K, Linnik MD. Evaluation of the safety of rituximab in combination with a tumor necrosis factor inhibitor and methotrexate in patients with active rheumatoid arthritis: results from a randomized controlled trial. Arthritis Rheum. 2011 Mar;63(3):622-32. doi: 10.1002/art.30194. PMID 21360491

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 17 sites in the United States.
Pre-assignment Details: After 24 weeks, participants continued post-treatment follow-up (PTFU) visits through Week 56, and entered a 48-week Safety Follow-Up (SFU). At any time between Week 24 and Week 40 of PTFU, eligible participants could enter the rituximab open label (OL) arm, and "restart" the 56-week treatment/follow-up schedule prior to the 48-week SFU.
Groups:
- Double-blind/Open Label Rituximab: The double-blind rituximab treatment group received rituximab 500 mg by intravenous (IV) infusion on Day 1 and Day 15. After 24 weeks (primary endpoint completion), participants continued post-treatment follow-up (PTFU) visits through Week 56, and entered a 48-week Safety Follow-Up (SFU). At any time between Week 24 and Week 40 of PTFU, eligible participants could enter the rituximab open label (OL) arm, and "restart" the 56-week treatment/follow-up schedule (rituximab 500 mg by IV infusion on Day 1 and Day 15) prior to the 48-week SFU.
- Double-blind Placebo/Open Label Rituximab: The double-blind placebo treatment group received saline solution IV on Day 1 and Day 15. After 24 weeks (primary endpoint completion), participants continued post-treatment follow-up (PTFU) visits through Week 56, and entered a 48-week Safety Follow-Up (SFU). At any time between Week 24 and Week 40 of PTFU, eligible participants could enter the rituximab open label (OL) arm, and "restart" the 56-week treatment/follow-up schedule (rituximab 500 mg by IV infusion on Day 1 and Day 15) prior to the 48-week SFU.
Period: Double-blind Phase
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Started | 36 (enrolled and randomized (2:1 scheme)) | 18
Safety Population | 33 (received treatment) | 18
Completed to Week 24 | 31 (received full course of rituximab therapy) | 18 (received full course of placebo therapy)
Completed to Week 56 | 8 | 3
Completed | 28 | 18
Not Completed | 8 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Failure to Return | 2 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Open Label Retreatment Phase
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Started | 22 | 16
Completed to Week 24 | 22 (received full course of open-label rituximab therapy) | 15 (received full course of open-label rituximab therapy)
Completed to Week 56 | 13 | 12
Completed | 13 | 12
Not Completed | 9 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Insufficient Therapeutic Response | 2 | 1
Not completed — Failure to Return | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Administrative/Other Reason | 2 | 0
Period: Safety Follow-up Phase
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Started | 22 | 17
Completed | 18 | 13
Not Completed | 4 | 4
Not completed — Failure to Return | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Administrative/Other Reason | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab | Total
Number analyzed (Participants) | 33 | 18 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (12.1) | 50.4 (11.4) | 50.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 17 | 45
  Male | 5 | 1 | 6
Years since rheumatoid arthritis (RA) diagnosis [Mean (Standard Deviation); unit: Years] | 10.3 (6.7) | 10.7 (7.5) | 10.5 (6.9)
Number of Prior Tumor Necrosis Factor (TNF) Inhibitors [Number; unit: participants]
  1 | 32 | 18 | 50
  2 | 1 | 0 | 1
C-Reactive Protein [Mean (Full Range); unit: mg/dL] | 0.97 [0.0 to 6.3] | 0.83 [0.1 to 3.3] | 0.92 [0.0 to 6.3]
Swollen and Tender Joints [Mean (Full Range); unit: Joint counts] — Total number of swollen joints evaluated was 66 and total number of tender joints evaluated was 68.
  Joint counts
    Swollen joints | 16.9 [5 to 43] | 14.2 [6 to 30] | 16.0 [5 to 43]
    Tender joints | 25.6 [5 to 56] | 22.8 [9 to 63] | 24.6 [5 to 63]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With at Least One Serious Infection Through Week 24
Description: An infection was considered serious if it required intravenous (IV) antibiotics or met the regulatory definition of a serious adverse event (SAE). An SAE was any event that resulted in death, resulted in a congenital anomaly in a child of a participant in the study, caused or prolonged an inpatient hospitalization, resulted in significant or persistent disability, or was considered by the investigator to be an important medical event that may have required intervention to prevent any of the above-listed outcomes.
Time Frame: Through Week 24
Population: The Safety Population consisted of all participants who received any part of an infusion of rituximab or placebo.
Measure: Number; unit: proportion of participants
Groups:
- Rituximab: The rituximab treatment group received rituximab 500 mg by intravenous infusion (IV) on Day 1 and Day 15. Prior to rituximab infusion, participants were premedicated with methylprednisolone 100 mg IV. Participants were also to receive a stable dose of folate ≥5 mg weekly.
- Placebo: The placebo treatment group received saline solution IV on Day 1 and Day 15. Prior to each infusion of placebo, participants were premedicated with methylprednisolone 100 mg IV. Participants were also to receive a stable dose of folate ≥5 mg weekly.
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 33 | 18
proportion of participants | 0.03 | 0.00

2. Secondary Outcome: Proportion of Participants Achieving an American College of Rheumatology 20 (ACR20) Response at Week 24
Description: An ACR20 response is defined as a 20% reduction in the number of both swollen and tender joints, and a 20% reduction in the score or results of at least 3 of the following 5 core set measurement tools: Patient and physician assessment of patient disease activity (DA) in previous 24 hours on a visual analog scale (VAS, no DA to maximum DA); patient assessment of pain in previous 24 hours on a VAS (none to unbearable); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Week 24
Population: The Safety Population consisted of all participants who received any part of an infusion of rituximab or placebo. Missing data were imputed using the nonresponder method, in which a participant with missing data at the visit being analyzed was considered a nonresponder.
Measure: Number; unit: proportion of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 33 | 18
proportion of participants | 0.30 | 0.17

3. Secondary Outcome: Proportion of Participants Achieving an American College of Rheumatology 50 (ACR50) Response at Week 24
Description: An ACR50 response is defined as a 50% reduction in the number of both swollen and tender joints, and a 50% reduction in the score or results of at least 3 of the following 5 core set measurement tools: Patient and physician assessment of patient disease activity (DA) in previous 24 hours on a visual analog scale (VAS, no DA to maximum DA); patient assessment of pain in previous 24 hours on a VAS (none to unbearable); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 33 | 18
proportion of participants | 0.12 | 0.06

4. Secondary Outcome: Proportion of Participants Achieving an American College of Rheumatology 70 (ACR70) Response at Week 24
Description: An ACR70 response is defined as a 70% reduction in the number of both swollen and tender joints, and a 70% reduction in the score or results of at least 3 of the following 5 core set measurement tools: Patient and physician assessment of patient disease activity (DA) in previous 24 hours on a visual analog scale (VAS, no DA to maximum DA); patient assessment of pain in previous 24 hours on a VAS (none to unbearable); Health Assessment Questionnaire-Disability Index (20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do); and C reactive protein or, if missing, erythrocyte sedimentation rate.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: proportion of participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 33 | 18
proportion of participants | 0.00 | 0.00

5. Primary Outcome: Number of Participants With Any Infections or Any Grade 3/4 Infections Through Week 24
Description: Infections were defined as adverse events that map to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) of "infections and infestations" and also included other infectious events that do not map to this SOC (e.g., cholecystitis, pleurisy, conjunctivitis, acne, tongue ulceration). Participants with multiple infections were calculated only once. The severity of all reported adverse events, including infections, was graded and reported according to the National Cancer Institute Common Terminology Criteria for Adverse Events. This scale defines the severity of an adverse event as follows: Grade 1 = a mild adverse event, Grade 2 = a moderate adverse event, Grade 3 = a severe adverse event, and Grade 4 = a life-threatening or disabling adverse event.
Time Frame: Through Week 24
Population: The Safety Population consisted of all participants who received any part of an infusion of rituximab or placebo.
Measure: Number; unit: participants
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Number analyzed (Participants) | 33 | 18
participants
  Any Infection | 18 | 11
  Any Grade 3/4 Infection | 3 | 0

6. Primary Outcome: Maximum Duration of Infections Through Week 24
Description: Infections were defined as adverse events that map to the Medical Dictionary for Regulatory Activities (MedDRA) system organ class (SOC) of "infections and infestations" and also included other infectious events that do not map to this SOC (e.g., cholecystitis, pleurisy, conjunctivitis, acne, tongue ulceration). For participants with multiple infections, only the infection with the longest duration was included in this analysis.
Time Frame: Week 24
Population: Participants in the Safety Population with at least 1 infection. The Safety Population consisted of all participants who received any part of an infusion of rituximab or placebo.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Number analyzed (Participants) | 18 | 11
days | 12.6 (9.6) [151.6 to 306.44] | 14.5 (5.2) [215.7 to 465.23]

7. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) Through Week 24
Description: An AE was any sign (including an abnormal laboratory result that the investigator determined to be clinically significant), symptom, or diagnosis/disease that is unfavorable or unintended, that was new, or if pre-existing, worsened in a participant and that did not necessarily have a causal relationship with the treatment. An SAE was any event that resulted in death, resulted in a congenital anomaly in a child of a participant in the study, caused or prolonged an inpatient hospitalization, resulted in significant or persistent disability, or was considered by the investigator to be an important medical event that may have required intervention to prevent any of the above-listed outcomes.
Time Frame: Through Week 24
Population: The Safety Population consisted of all participants who received any part of an infusion of rituximab or placebo.
Measure: Number; unit: participants
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Number analyzed (Participants) | 33 | 18
participants
  Any AE | 31 | 15
  Any SAE | 2 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Immunological and Laboratory Assessment Findings
Description: The following immunological assessments were conducted: autoantibody concentrations for RF, anti-cyclic-citrullinated peptide (CCP) antibody concentrations, quantitative immunoglobulin levels, and lymphocyte assessments of T- and B-cell populations, determined using whole blood expanded fluorescent-activated cell sorter (FACS) analysis. The following laboratory assessments were performed: hemoglobin, hematocrit, red blood cells (RBC), white blood cells (WBC) with differential, and platelet counts; aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total protein, albumin, total bilirubin, blood urea nitrogen (BUN), uric acid, creatinine, random glucose, potassium, sodium, chloride, calcium, and phosphorous; blood, protein, and glucose (microscopic examination, if abnormal and applicable).
Time Frame: Through Week 24
Population: The Safety Population consisted of all participants who received any part of an infusion of rituximab or placebo.
Measure: Number; unit: participants
Arm/Group | Double-blind/Open Label Rituximab | Double-blind Placebo/Open Label Rituximab
Number analyzed (Participants) | 33 | 18
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: For Double-Blind Rituximab and Double-Blind Placebo reporting groups, nonserious AE data and SAE data are presented through the Week 24 treatment phase (primary endpoint completion). See Additional Description (below) for Cumulative Rituximab time frame.
Description: For Cumulative Rituximab reporting group, nonserious AEs were captured only through Week 56. Serious adverse events (SAEs) were captured during treatment and post-treatment periods, through the safety follow-up (SFU) period (48 weeks) and the extended safety follow-up (ESFU; 1760 days).
Groups:
- Double-Blind Rituximab: The rituximab treatment group received rituximab 500 mg by intravenous infusion (IV) on Day 1 and Day 15. Prior to rituximab infusion, participants were premedicated with methylprednisolone 100 mg IV. Participants were also to receive a stable dose of folate ≥5 mg weekly.
- Double-Blind Placebo: The placebo treatment group received saline solution IV on Day 1 and Day 15. Prior to each infusion of placebo, participants were premedicated with methylprednisolone 100 mg IV. Participants were also to receive a stable dose of folate ≥5 mg weekly.
- Cumulative Rituximab: The cumulative rituximab treatment group included all participants who received rituximab at any time during the study, including participants who received rituximab in the double-blind period and did not participate in the OL period, those who received placebo in the double-blind period and rituximab in the OL, and those who received rituximab in the double-blind and OL periods. Prior to rituximab infusion, participants were premedicated with methylprednisolone 100 mg IV. Participants were also to receive a stable dose of folate ≥5 mg weekly.
Arm/Group | Double-Blind Rituximab | Double-Blind Placebo | Cumulative Rituximab
Serious Adverse Events (participants affected / at risk) | 2/33 | 0/18 | 8/49
Other Adverse Events (participants affected / at risk) | 31/33 | 15/18 | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Rituximab (N=33) | Double-Blind Placebo (N=18) | Cumulative Rituximab (N=49)
Coronary Artery Occlusion (Cardiac disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Arthritis Infective (Infections and infestations) | 0 | 0 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Rituximab (N=33) | Double-Blind Placebo (N=18) | Cumulative Rituximab (N=49)
Insomnia (Psychiatric disorders) | 3 | 0 | 4
Edema peripheral (General disorders) | 3 | 2 | 5
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Headache (Nervous system disorders) | 3 | 2 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 5 | 15
Asthenia (General disorders) | 2 | 1 | 2
Flushing (Vascular disorders) | 2 | 0 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 5
Dizziness (Nervous system disorders) | 3 | 1 | 4
Anxiety (Psychiatric disorders) | 3 | 0 | 4
Infusion-related reaction (General disorders) | 2 | 1 | 5
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4
Fatigue (General disorders) | 4 | 0 | 5
Blood glucose increased (Investigations) | 2 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 14
Vaginal mycosis (Infections and infestations) | 2 | 1 | 4
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 5 | 2 | 7
Sinusitis (Infections and infestations) | 3 | 3 | 14
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6
Vomiting (Gastrointestinal disorders) | 3 | 0 | 5
Bronchitis (Infections and infestations) | 1 | 1 | 5
Gastroenteritis (Infections and infestations) | 1 | 1 | 2
Herpes Simplex (Infections and infestations) | 0 | 1 | 0
Infected Insect Bite (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 2
Postoperative Infection (Infections and infestations) | 1 | 0 | 1
Tooth Abscess (Infections and infestations) | 1 | 0 | 3
Tooth Infection (Infections and infestations) | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Seasonal Allergy (Immune system disorders) | 1 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 1
Stress (Psychiatric disorders) | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Restless Legs Syndrome (Nervous system disorders) | 1 | 0 | 1
Eyelid Oedema (Eye disorders) | 1 | 0 | 1
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Ear Pruritus (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
Raynaud's Phenomenon (Vascular disorders) | 0 | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Abdominal Adhesions (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 2
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 3
Rectocele (Gastrointestinal disorders) | 1 | 0 | 1
Tooth Fracture (Gastrointestinal disorders) | 0 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cystocele (Renal and urinary disorders) | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Genital Pruritus Female (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1
Chest Pain (General disorders) | 1 | 0 | 1
Oedema (General disorders) | 0 | 1 | 0
Venipuncture Site Inflammation (General disorders) | 1 | 0 | 1
Bacteria Sputum Identified (Investigations) | 0 | 1 | 0
Blood Calcium Increased (Investigations) | 1 | 0 | 1
Blood Phosphorus Decreased (Investigations) | 1 | 0 | 1
Heart Rate Increased (Investigations) | 0 | 1 | 0
Lymphocyte Count Increased (Investigations) | 1 | 0 | 1
Monocyte Count Increased (Investigations) | 1 | 0 | 1
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 3
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin Injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 3
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 3
Acute Sinusitis (Infections and infestations) | 0 | 0 | 1
Arthritis Infective (Infections and infestations) | 0 | 0 | 1
Bronchitis Acute (Infections and infestations) | 0 | 0 | 1
Dental Caries (Infections and infestations) | 0 | 0 | 1
Dermatophytosis (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Dry Socket (Infections and infestations) | 0 | 0 | 1
Ear Infection (Infections and infestations) | 0 | 0 | 1
Eye Infection (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1
Oral Fungal Infection (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Tinea Infection (Infections and infestations) | 0 | 0 | 1
Tinea Pedis (Infections and infestations) | 0 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 1
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Benign Neoplasm Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 2
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes Mellitus Non-Insulin-Dependent (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 1
Neuropathy (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 3
Dry Eye (Eye disorders) | 0 | 0 | 1
Coronary Artery Atherosclerosis (Cardiac disorders) | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 0 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal Polyp (Gastrointestinal disorders) | 0 | 0 | 1
Reflux Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Salivary Gland Calculus (Gastrointestinal disorders) | 0 | 0 | 1
Swollen Tongue (Gastrointestinal disorders) | 0 | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Heat Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Idiopathic Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sebaceous Hyperplasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Rheumatoid Nodule (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Ganglion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Dermoid Cyst (Congenital, familial and genetic disorders) | 0 | 0 | 1
Localised Oedema (General disorders) | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1
Mean Cell Volume Increased (Investigations) | 0 | 0 | 1
Platelet Count Increased (Investigations) | 0 | 0 | 1
Weight Increased (Investigations) | 0 | 0 | 1
Incision Site Complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Sponsor made a business decision to terminate study on 28 July 2011, after completion of the primary endpoint and during the long-term extension phase. One participant was still in extended safety follow-up and was referred for appropriate care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.